CLINICAL TRIAL: NCT03109509
Title: Pokémon Go Modestly Increases Time Spent Active Among Healthy Adults
Brief Title: Testing the Efficacy of Pokemon Go for Increasing Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lucas Carr, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201607768; 5K25HL122305 (NIH)
Record Dates: First submitted 2017-04-05; First posted 2017-04-12 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Two-group, randomized controlled trial.
Who Masked: Investigator
Masking Description: Research team was blinded to participant group assignment until data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit-only Group (Active Comparator): Participants randomized to the FB group were provided a Fitbit Zip activity monitor and were instructed on how to wear the monitor, how to pair the activity monitor to their smartphone, and asked to provide our team consent to access their Fitbit data through Fitbit's Application Programming Interface (API)
  Interventions: Behavioral: Fitbit Only
- Fitbit + Pokémon Go Group (Experimental): Participants randomized to the FB+P group received the same Fitbit Zip activity monitor and text message reminders as the FB group. This group was also shown how to download the Pokémon Go application to their smartphone and were provided brief instructions on how to play the game. Participants were instructed to simply explore the game and play it at their leisure. Participants were not provided any specific goals related to game play or physical activity in general.
  Interventions: Behavioral: Fitbit + Pokemon Go

INTERVENTIONS:
Behavioral: Fitbit + Pokemon Go — Participants received a Fitbit Zip to wear daily for 8 weeks. Participants also received access to the Pokemon Go game.
  Arms: Fitbit + Pokémon Go Group
Behavioral: Fitbit Only — Participants received a Fitbit Zip to wear daily for 8 weeks.
  Arms: Fitbit-only Group

SUMMARY:
Historically, increasing activity was synonymous with exercise; however, it is now thought that even much more modest activity levels (e.g., simply walking) or merely decreasing the proportion of sedentary time may be sufficient to decrease future morbidity and mortality. Some interventions designed to increase activity have shown promise; others have been less successful. But even promising interventions are often difficult to generalize to real-life clinical settings. One barrier to monitoring the effectiveness of interventions has been the lack of availability of accurate, reliable and inexpensive personal activity monitoring equipment. The availability of inexpensive pedometers, and, more recently, low cost triaxial accelerometers, has now made it much easier to monitor activity levels and provide feedback to users. These devices are ideal for capturing activity associated with walking, the most popular and acceptable form of exercise, but only if patients actually wear them. Thus, there is a need to develop pragmatic approaches that encourage patients to not only wear these monitoring devices, but also motivate them to increase their activity.

In recent years, games have been used in a variety of settings to motivate and change behavior. Games not only provide performance feedback to patients, but also provide incentives for achieving goals in a context that is fun, intrinsically rewarding, and easy to understand. Successful games effectively exploit motivating social factors (e.g., competition, peer support, and entertainment) to maintain interest and engage participants. Steps are counted using a commercially available triaxial accelerometer (e.g., a FitBit). Pokemon Go is an augmented reality game that encourages players to go outside to search for Pokemon creatures.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age, healthy adults, own smart phone, have access to the Internet, fluent in English, no contraindications to physical activity, not pregnant or planning to become pregnant, had not previously played Pokemon Go game

Exclusion Criteria:

* <18 year or older than 80 years of age, did not own smart phone, did not have access to the Internet, not fluent in English, any contraindications to physical activity, pregnant or planning to become pregnant in next 2 months, had previously played Pokemon Go game

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Average daily steps | Eight weeks
  Daily steps measured by Fitbit Zip

IPD SHARING:
Plan to Share IPD: No
No plan to share individual data with other researchers.